CLINICAL TRIAL: NCT01758198
Title: A Phase 4, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Abatacept in Combination Therapy With Methotrexate vs. Methotrexate Alone in Subjects With Active Rheumatoid Arthritis and Inadequate Response to Methotrexate
Brief Title: Abatacept Post-marketing Clinical Study in Japan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM101-338
Record Dates: First submitted 2012-12-19; First posted 2013-01-01 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: Abatacept + Methotrexate (MTX) (Experimental): Abatacept 10 mg/kg solution intravenous (IV) infusion, once monthly for 12 months
  Methotrexate ≥6 mg/week for 12 months
  Interventions: Biological: Abatacept; Drug: Methotrexate
- Group 2: Placebo matching with Abatacept + Methotrexate (Placebo Comparator): Placebo matching with Abatacept 0 mg/kg solution, intravenous (IV) infusion once monthly for 12 months
  Methotrexate ≥6 mg/week for 12 months
  Interventions: Drug: Placebo matching with Abatacept; Drug: Methotrexate

INTERVENTIONS:
Biological: Abatacept
  Other Names: BMS-188667 (Orencia)
  Arms: Group 1: Abatacept + Methotrexate (MTX)
Drug: Placebo matching with Abatacept
  Arms: Group 2: Placebo matching with Abatacept + Methotrexate
Drug: Methotrexate

SUMMARY:
The purpose of this study is to compare the clinical efficacy including joint damage progression and safety of Abatacept plus Methotrexate (MTX) to placebo plus MTX.

ELIGIBILITY:
Inclusion Criteria:

* MTX inadequate responder
* Biologic Naïve
* Functional class I, II or III
* ≥6 swollen and ≥6 tender joints
* C-reactive protein (CRP) ≥2.0mg/dl or erythrocyte sedimentation rate (ESR) ≥28 mm/hr
* Anti-cyclic citrullinated peptide (CCP) antibody positive
* Have erosion

Exclusion Criteria:

* Any other rheumatic disease
* Active angiitis on main organs excluding rheumatoid nodule

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2013-04-11 (Actual); Primary Completion 2016-12-26 (Actual); Study Completion 2016-12-26 (Actual)

PRIMARY OUTCOMES:
American College of Rheumatology (ACR) 20% response rate | 4 months (week 16)
Change from baseline in Total Sharp Score (TSS) using the Modified van der Heijde Sharp (vdH-S) method to 6 months (Week 24) | Baseline (Day 1), 6 months (Week 24)

SECONDARY OUTCOMES:
Change from baseline in Disease Activity Score-28 (DAS28)-CRP to 4 months (Week16) | Baseline (Day 1), 4 months (Week 16)
Non-progressors rate for the structural damage | Baseline (Day 1), 6 months (Week 24)
  The non-progressors rate is defined as the proportion of subjects meeting the change from baseline in the TSS at 6 months less than or equal to the smallest detectable difference (SDD) and/or the smallest detectable change (SDC)
ACR 50 response rates | 4 months (Week16)
ACR 70 response rates | 4 months (Week16)
Safety and tolerability will be measured based on clinical Adverse Events, vital signs, and laboratory abnormalities | 12 months (Week52)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (55):
- Japan (55):
  - Local Institution, Kamogawa, Chiba
  - Local Institution, Kasamatsu-town, Gifu
  - Local Institution, Kakogawa, Hyōgo
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Kurashiki, Okayama-ken
  - Local Institution, Izumisano, Osaka
  - Local Institution, Fujieda, Shizuoka
  - Local Institution, Toyama, Toyama
  - Local Institution, Shimonoseki, Yamaguchi
  - Local Institution, Asahi
  - Local Institution, Fuchū
  - Local institution, Fukuoka
  - Local Institution, Fukuoka
  - Local institution, Funabashi
  - Local Institution, Hakodate
  - Local Institution, Hiroshima
  - Local Institution, Hitachi
  - Local institution, Hokkaido
  - Local Institution, Iizuka
  - Local Institution, Kagoshima
  - Local Institution, Kanazawa
  - Local Institution, Kasama
  - Local Institution, Katō
  - Local Institution, Kitakyushu
  - Local Institution, Kitamoto
  - Local institution, Kobe
  - Local Institution, Kochi
  - Local Institution, Kōshi
  - Local institution, Kumamoto
  - Local Institution, Matsumoto
  - Local Institution, Nagano
  - Local Institution, Nagaoka
  - Local Institution, Nagasaki
  - Local Institution, Nagoya
  - Local Institution, Narashino
  - Local Institution, Narita
  - Local Institution, Okayama
  - Local institution, Osaka
  - Local institution, Ōme
  - Local Institution, Ōsaki
  - Local institution, Sapporo
  - Local Institution, Sapporo
  - Local Institution, Sasebo
  - Local Institution, Sayama
  - Local Institution, Sendai
  - Local Institution, Shizuoka
  - Local Institution, Takaoka
  - Local Institution, Takasaki
  - Local institution, Tokyo
  - Local Institution, Tokyo
  - Local Institution, Tomakomai
  - Local Institution, Toyama
  - Local Institution, Utsunomiya
  - Local institution, Yokohama
  - Local Institution, Yotsukaidō

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx